CLINICAL TRIAL: NCT02125058
Title: Randomized Controlled Trial for the Cosmetic Result of Intracutaneous Versus Transcutaneous Sutures After Dermatologic Surgery in the Face
Brief Title: Intracutaneous Versus Transcutaneous Sutures in the Face (IC vs TC Sutures)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL46056.068.13
Record Dates: First submitted 2014-01-15; First posted 2014-04-29 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2015-04

CONDITIONS: Skin Tumour; Surgery
Keywords: intracutaneous sutures; transcutaneous sutures; dermatological surgery; facial area
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous sutures (Other): Transcutaneous sutures
  Interventions: Procedure: Transcutaneous sutures
- Intracutaneous sutures (Other): Intracutaneous sutures
  Interventions: Procedure: Intracutaneous sutures

INTERVENTIONS:
Procedure: Transcutaneous sutures — Conventional excision followed by subcutaneous sutrues and transcutaneous sutures
  Arms: Transcutaneous sutures
Procedure: Intracutaneous sutures — Conventional excision followed by subcutaneous sutrues and intracutaneous sutures
  Arms: Intracutaneous sutures

SUMMARY:
Rationale:

Skin cancer is common in Caucasians and often exists on sun-exposed areas, such as the face. Treatment of choice is mostly excision and result in an irreversible scar. As the incidence of skin cancer is rising, also among young people, it is important to obtain a good cosmetic outcome after treatment. It is believed that the type of closure of the wound after excision can influence the cosmetic result. Currently, primary closure of the excision can occur by transcutaneous (TC) or intracutaneous (IC) suturing. Both techniques are widely used among dermatologists and plastic surgeons and the choice is mainly dependent on the preference of the physician. Research comparing the cosmetic result of both techniques in the craniofacial area is lacking.

Objective:

Evaluation of the cosmetic result of transcutaneous sutures versus intracutaneous sutures in the craniofacial area.

Study design:

A randomized controlled single-blinded multi-center trial.

Study population:

Patients older than 18 years, with craniofacial skin tumor receiving surgery followed by primary closure at the department of Dermatology and Plastic Surgery of the Maastricht University Medical Centre, the department of Dermatology of Catharina hospital Eindhoven and the department of Plastic surgery of Orbis Medical Centre Sittard.

Intervention:

Excision of the tumor followed by IC sutures or TC sutures

Main study endpoints:

Cosmetic result measured on the Patient and Observer Scar Assessment Scale (POSAS) by the patient and the researcher 12 months after surgery.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

All patients who participate have an indication for excision and will be assigned to one of the suture techniques. Both techniques are widely used in the regular patient care. Therefore, no extra risks are associated with it.

Patients will be asked to visit the hospital 3 months and 1 year following treatment, at which point a questionnaire will be filled in and the redness of the scar will be measured by means of non-invasive techniques. In addition, patients will be asked to apply a sunscreen on the scar daily during the first three months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older with a skin tumour of minimal 5mm in diameter in the craniofacial area requiring an excision followed by primary closure will be included. If a patient has more than one lesion, the largest lesion that can be closed primarily will be included as a maximum of one tumour per patient will be studied.

Exclusion Criteria:

* Patients with skin lesions on the ears, nose, mucosal part of the lips or eyelids as patients suited for excision but where a transplantation, flap or secondary granulation is necessary for reconstruction of the defect will be excluded. Patients not capable of informed consent will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The study aims to evaluate the cosmetic outcome 12 months post-treatment of IC compared to TC sutures after excision of a skin tumor in the face. Cosmetic result after surgery in the face | after 1 year
  The study aims to evaluate the cosmetic outcome 12 months post-treatment of IC compared to TC sutures after excision of a skin tumor in the face.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomeng Liu, drs., Principal Investigator — Maastricht University Hospital
Locations (3):
- Netherlands (3):
  - Maastricht University Hospital, Maastricht, Limburg
  - Orbis Medical Center, Sittard, Limburg
  - Catharina Hospital, Eindhoven, North Brabant